CLINICAL TRIAL: NCT02629263
Title: The Effect of Viscous Fibre on Glycemic Control in Individuals With Diabetes
Brief Title: The Effect of Viscous Fiber on Glycemic Control in Individuals With Diabetes
Acronym: VF&GC
Status: Completed | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: Viscous Fiber and GC
Record Dates: First submitted 2015-11-27; First posted 2015-12-14 (Estimated); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Viscous Fiber — Meta- analysis of Randomized Controlled Trials

SUMMARY:
Purpose of Study (The Effect of Viscous Fiber on Glycemic Control (VF & GC) in Individuals with Diabetes Mellitus.

According to the World Health Organization, about 347 million individuals are living with diabetes. (http://www.who.int/features/factfiles/diabetes/facts/en/, accessed on Nov. 23, 2015). Over the last decades, dietary fibers, namely dietary viscous fibers, have emerged as a nutrition component that may improve the postprandial glycemic response and hence aid in long term diabetes management. It is believed that supplementation with viscous fibers can control blood glucose by increasing viscosity of the gastric digesta, hence delaying gastric emptying and retarding entry of glucose into the bloodstream to result in a diminished postprandial rise in blood glucose. (Chutkan et al., 2012).

Currently, the evidence of the relationship between viscous fibers and diabetes is mixed. The systematic review method depends on combining data from many small studies in order to get a pooled estimate of the true effect. The purpose of this study is to conduct a systematic review and meta-analysis of randomized controlled trials (RCTs) investigating the fasting glycemic and insulinemic effect of viscous fiber supplementation. We hope the findings of this study will play a key role in developing the nutritional guidelines for individuals with diabetes mellitus.

DETAILED DESCRIPTION:
Background: Diet high in total dietary fiber content has been recommended for individuals with diabetes mellitus. However, the effect of supplementing diet with viscous fiber such as guar gum, beta glucan, psyllium, konjac, or other viscous fibers on glycemic and insulinemic outcomes in individuals with diabetes mellitus is still controversial.

Objective: To improve the evidence-based guidelines/ recommendations for diabetes mellitus, we will conduct a systematic review and meta-analysis on the effect of viscous fiber supplementation on glycemic control endpoints in individuals with diabetes mellitus.

Design: Cochrane handbook for systematic review of interventions will be used for planning and conducting this meta-analysis. The reporting will follow the Preferred Reporting Items for Systematic Reviews and Meta-analyses (PRISMA) guidelines.

Data sources: MEDLINE, EMBASE, the Cochrane Central Register of Controlled Trials will be searched using appropriate pre-determined search terms.

Study selection: All the included trials must be randomized, controlled, with duration of ≥ 3 weeks investigating the effect of supplementing diet with viscous fiber on glycemic control outcomes in individuals with diabetes mellitus. Acute studies, non-randomized, not appropriately controlled studies will be excluded. Both isocaloric and non-isocaloric will be included.

Data extraction: Two independent reviewers will extract information about fiber type, sample size, subject characteristics, dose, follow-up, composition of the background diets, and statistical analyses. Mean±SEM values will be extracted for all outcomes. Standard computation and imputation will be used to derive all missing variance data. Risk of bias and study quality will be assessed using the Cochrane Risk of Bias Tool and the Grading of Recommendations Assessment, Development and Evaluation (GRADE), respectively.

Outcome: This meta-analysis will assess a set of outcomes related to glycemic control in individuals with diabetes mellitus. These outcomes are: (1) glycated hemoglobin A1c (HbA1c), (2) fasting glucose (FG), (3) fasting insulin (FI), (4) fructosmine, and (5) Homeostasis model assessment of insulin resistance (HOMA-IR).

Data synthesis: Pooled analysis will be conducted using the Generic Inverse Variance method. Rand-effects models will be used even in the absence of statistical significant between-study heterogeneity because they yield more conservative summary effect estimates in the presence of residual heterogeneity. Heterogeneity will be assessed using Cochran's Q test and quantified by the I2 statistic. Sensitivity and subgroup analyses will be used to explore sources of heterogeneity. A prioir subgroup analyses include study design, does, fiber type, follow-up (duration), baseline values, study quality, food matrix, and composition of the background diet. The significance of subgroup analyses will be assessed using meta-regression analyses. Publication bias will be assessed using the inspection of funnel plots and application of Egger's and Begg's tests.

Knowledge translation plan: Results will be shared through traditional, national, and international scientific meetings and they will be submitted to high impact factor journals for publication.

Significance: We hope the results of this study will play a role in improving the guidelines/ recommendations for individuals with diabetes mellitus by raising the awareness towards viscous fiber consumption among health providers, patients, and industry. Hopefully, this study will aid in guiding future research in the dietary fiber field.

ELIGIBILITY:
Inclusion Criteria:

* Randomized Controlled Trials
* Parallel or Crossover Design
* Duration: ≥ 3 weeks
* Food/ Supplements.
* Soluble Fibers include: B-Glucan, Guar Gum, Konjac, Pectin, Psyllium.
* Diabetes Biomarkers include: Fasting Blood Glucose, Fasting Insulin, Fructosamine, and HbA1c.

Exclusion Criteria:

--------

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study includes all population types.
Sampling Method: Probability Sample
Enrollment: 1394 (Actual)
Dates: Start 2015-09; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
HbA1c (%) | 3 weeks

SECONDARY OUTCOMES:
Fasting Blood Glucose (mmol/l) | ≥ 3 weeks
Fasting Blood Insulin (pmol/l) | ≥ 3 weeks
Fructosamine (mmol/l) | ≥ 3 weeks
HOMA-IR (mU/mmol/l) | ≥ 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, PhD, Principal Investigator — St.Michael Hospital
Locations (1):
- Clinical Nutrition and Risk Factor Modification Centre, Toronto, Ontario, Canada